CLINICAL TRIAL: NCT01456975
Title: Reimplantation Procedure for Surgical Treatment of Ascending Aorta Aneurism With Concomitant Aortic Valve Insufficiency
Brief Title: Extravalvular Procedure for Surgical Treatment of Ascending Aorta Aneurism
Acronym: EPSTAAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EVAPRO
Record Dates: First submitted 2011-09-27; First posted 2011-10-21 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Ascending Aorta Aneurism; Aortic Insufficiency
Keywords: Ascending aorta aneurism; Aortic insufficiency
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Valsalva (Experimental): Reimplantation procedure using Valsalva prosthesis
  Interventions: Procedure: Aortic valve reimplantation using Valsalva prosthesis

INTERVENTIONS:
Procedure: Aortic valve reimplantation using Valsalva prosthesis — Aortic valve reimplantation (David procedure)using Valsalva prosthesis
  Other Names: Gelweave Vascutek Valsalva

SUMMARY:
The investigators expect that the using of prothesis with sinuses has more benefits for long term competence and condition of aortic valve than the using of straight prothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Aortic insufficiency 2+
2. Ascending aorta size more than 5 cm
3. Ascending aorta size more than 4,5 cm (Marfan syndrome)
4. Good conditions of aortic cusps

Exclusion Criteria:

1. Aortic annulus more than 30 mm
2. Aortic cusps destruction
3. Critical aortic cusps elongation
4. Aortic root dissection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-01; Primary Completion 2012-12 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
all causes of aortic valve replacement | before discharging (average of 2 weeks after surgery)
  Aortic insufficiency (AI) measured by echocardiography. If AI more than 2+, aortic valve replacement performed

SECONDARY OUTCOMES:
all causes of death after procedure | 6, 12, 24,36,48,60,72, 84, 96 months after procedure
  Aortic insufficiency (AI) measured by echocardiography. If AI more than 2+, aortic valve replacement performed

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry A. Sirota, Novosibirsk, Russia